CLINICAL TRIAL: NCT05649787
Title: Effects of a Supervised Training Program on Functional Capacity in Patients With Heart Failure and Preserved Ejection Function and Chronotropic Incompetence
Brief Title: Effects of a Supervised Training Program on Functional Capacity in Patients With HFpEF and Chronotropic Incompetence
Acronym: Training-HR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación para la Investigación del Hospital Clínico de Valencia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Training-HR
Record Dates: First submitted 2022-11-22; First posted 2022-12-14 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Heart Failure With Preserved Ejection Fraction; Chronotropic Incompetence
Keywords: Heart Failure with Preserved Ejection Fraction; Chronotropic incompetence; Functional capacity

STUDY DESIGN:
Intervention Model Description: This is a prospective study, blinded for the evaluator, randomized (1:1:1:1) to receive standard management alone or combined with a program of training (aerobic alone or combined with strength exercises) that will be carried out in a single centre.
Who Masked: Investigator
Masking Description: Blinded only for the evaluator of primary and secondary endpoints
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Usual care (No Intervention): Patients allocated to this arm will receive the usual care plus explicit recommendations for home-based aerobic and strength training.
- Supervised aerobic training (Active Comparator): Patients allocated to this arm will receive the usual care plus supervised aerobic training
  Interventions: Behavioral: Supervised aerobic training
- Supervised aerobic plus low to moderate-intensity strenght training (Active Comparator): Patients allocated to this arm will receive the usual care plus supervised aerobic and low to moderate-intensity strength training
  Interventions: Behavioral: Supervised aerobic training; Behavioral: Supervised aerobic plus low to moderate-intensity strength training
- Supervised aerobic plus moderate to high-intensity strenght training (Active Comparator): Patients allocated to this arm will receive the usual care plus supervised aerobic and moderate to high-intensity strength training.
  Interventions: Behavioral: Supervised aerobic training; Behavioral: Supervised aerobic plus moderate to high-intensity strength training

INTERVENTIONS:
Behavioral: Supervised aerobic training — Supervised moderate to high-intensity interval aerobic training
  Arms: Supervised aerobic plus low to moderate-intensity strenght training; Supervised aerobic plus moderate to high-intensity strenght training; Supervised aerobic training
Behavioral: Supervised aerobic plus low to moderate-intensity strength training — Supervised moderate to high-intensity interval aerobic training plus low to moderate-intensity strength training
  Arms: Supervised aerobic plus low to moderate-intensity strenght training
Behavioral: Supervised aerobic plus moderate to high-intensity strength training — Supervised moderate to high-intensity interval aerobic training plus moderate to high-intensity strength training
  Arms: Supervised aerobic plus moderate to high-intensity strenght training

SUMMARY:
This is a prospective study, blinded for the evaluator, randomized (1:1:1:1) to receive standard management alone or combined with a program of training (aerobic alone or combined with strength exercises) that will be carried out in a single centre. After randomization, patients will be clinically evaluated. The primary endpoint (peakVO2) will be assessed by cardiopulmonary exercise testing (CPET) at 12 weeks. Patients with heart failure with preserved ejection fraction, functional class NYHA II-III, and chronotropic incompetence criteria will be enrolled. A sample size estimation [alfa: 0.05, power: 80%, a 15% loss rate, and at least a delta change of mean peakVO2: +2,4 mL/kg/min (SD±2)] of 80 patients (20 per arm) would be necessary to test our hypothesis.

DETAILED DESCRIPTION:
Heart failure with preserved ejection fraction (HFpEF) is a highly prevalent clinical entity that predominantly affects women >60 years old, whose incidence has increased in the last decade and has a complex and multifactorial pathophysiology. Chronotropic incompetence (CrI) has emerged as a crucial mechanism, particularly in patients older than 60 years, and is associated with more significant functional impairment. Supervised training programs in patients with heart failure and reduced ejection fraction and CrI have improved functional capacity and chronotropic response. However, we do not have evidence about the effects of a supervised training program on patients with HFpEF and CrI. This work aims to evaluate the effect of a supervised exercise program for 12 weeks in patients with HFpEF and CrI on peak oxygen consumption (peakVO2) and chronotropic response.

This is a prospective study, blinded for the evaluator, randomized (1:1:1:1) to receive standard management alone or combined with a program of training (aerobic alone or combined with strength exercises) that will be carried out in a single centre. After randomization, patients will be clinically evaluated. The primary endpoint (peakVO2) will be assessed by cardiopulmonary exercise testing (CPET) at 12 weeks. Patients with HFpEF, functional class NYHA II-III, and CrI criteria will be enrolled. A sample size estimation [alfa: 0.05, power: 80%, a 15% loss rate, and at least a delta change of mean peakVO2: +2,4 mL/kg/min (SD±2)] of 80 patients (20 per arm) would be necessary to test our hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with heart failure with preserved ejection fraction according to 2021 ESC guidelines for Heart Failure.
* N-terminal pro-B-type natriuretic peptide (NT-proBNP) >125 pg/mL in the last month
* Stable symptomatic heart failure patients (New York Heart Association functional class II-III/IV) during the last month
* Age ≥ 60 years old.
* Blunted heart rate (HR) response during a maximal cardiopulmonary exercise testing (CPET), defined as a chronotropic index <0.62 if previous treatment with Beta-blockers or chronotropic index <0.80 in patients without beta-blockers. Chronotropic index= [HRpeak exercise - HRrest] / [220 - age - HRrest]

Exclusion Criteria:

* Inability to perform a valid baseline cardiopulmonary exercise test
* Cardiac pacemaker
* Significant primary moderate-to-severe valve disease
* Effort angina or signs of ischemia during CPET
* Primary cardiomyopathies
* Cardiac transplantation
* Any other comorbidity with a life expectancy of less than one year

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-01-18 (Actual); Primary Completion 2024-11-18 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Peak oxygen consumption | Peak oxygen consumption will be evaluated at first visit and after 3 months. We will evaluate peak oxygen consumption change from baseline.
  Maximal functional capacity will be evaluated using incremental and symptom-limited cardiopulmonary exercise testing on a bicycle ergometer, beginning with a workload of 10 W and increasing gradually in a ramp protocol at 10-W increments every 1 minute. We define maximal functional capacity as when the patient stops pedalling because of symptoms and the respiratory exchange ratio (RER) was >1. During exercise, patients will be monitored with 12-lead electrocardiogram and blood pressure measurements every 2 minutes. Gas exchange data and cardiopulmonary variables were averages of values taken every 10 seconds. Peak oxygen consumption (PeakVO2) was defined as the highest value of VO2 during the last 20 seconds of exercise.
  Primary outcome: changes in peak oxygen consumption between and within groups at 12-week Unit of measure of peak oxygen consumption: mL/kg/min

SECONDARY OUTCOMES:
Chronotropic response | Chronotropic index will be evaluated at first visit and after 3 months. We will evaluate chronotropic index change from baseline.
  Heart rate (HR) response during the maximal cardiopulmonary exercise testing will be evaluated following the chronotropic index (CIx) formula. The chronotropic index is evaluated by the following formula, including heart rate at peak effort, heart rate at rest and age. Chronotropic index: (peak heart rate-rest heart rate)/ [220-age-rest heart rate)].
  Secondary outcome: changes in chronotropic response in between and within groups at 12-week Heart rate unit: beats per minute Age unit: years The chronotropic index has no units of measure.
Kansas City Cardiomyopathy Questionnaire Scales | The Kansas City Cardiomyopathy Questionnaire will be evaluated at first visit and after 3 months. We will evaluate the Kansas City Cardiomyopathy Questionnaire change from baseline.
  The Kansas City Cardiomyopathy Questionnaire includes 23 items that map to 7 domains: symptom frequency, symptom burden, symptom stability, physical limitations, social limitations, quality of life, and self-efficacy (the patient's understanding of how to manage their heart failure). All Kansas City Cardiomyopathy Questionnaire domains are scaled from 0 to 100, where scores represent health status as follows: 0 to 24, very poor to poor; 25 to 49, poor to fair; 50 to 74, fair to good; and 75 to 100, good to excellent.
  A change of 5 points is considered to be a small but clinically important change, whereas changes of 10 and 20 points are considered moderate-to-large and large-to-very-large clinical changes.

CONTACTS AND LOCATIONS:
Overall Officials: Patricia Palau, MD, PhD, Principal Investigator — Instituto de Investigacion Sanitaria INCLIVA
Locations (1):
- INCLIVA, Valencia, Spain

REFERENCES:
- [Derived] Palau P, de Amo I, Nunez G, Flor C, de la Espriella R, Garcia-Conejo C, Berlanga-Tovar SE, Casana-Granell J, Calatayud J, Dominguez E, Sanchis-Gomar F, Meyer M, Sanchis J, Nunez J, Lopez L. Effect of exercise training in patients with chronotropic incompetence and heart failure with preserved ejection fraction: the TRAINING-HR randomized clinical trial. Eur J Prev Cardiol. 2026 Feb 3;33(2):265-275. doi: 10.1093/eurjpc/zwaf269. Erratum In: Eur J Prev Cardiol. 2025 Dec 30:zwaf781. doi: 10.1093/eurjpc/zwaf781. PMID 40294211
- [Derived] Palau P, Nunez J, Dominguez E, de la Espriella R, Nunez G, Flor C, de Amo I, Casana J, Calatayud J, Ortega L, Marin P, Sanchis J, Sanchis-Gomar F, Lopez L. Effect of exercise training in patients with chronotropic incompetence and heart failure with preserved ejection fraction: Training-HR study protocol. Curr Probl Cardiol. 2024 Dec;49(12):102839. doi: 10.1016/j.cpcardiol.2024.102839. Epub 2024 Sep 4. PMID 39242065